CLINICAL TRIAL: NCT06300502
Title: Assessing the Efficacy of Repeat, Monthly Treatments of Cutaneous Neurofibromas (cNFs)
Brief Title: Assessing the Efficacy of Repeat, Monthly Treatments of Deoxycholate for NF1 Associated Cutaneous Neurofibromas (cNFs)
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Johns Hopkins University (Other); Neurofibromatosis Therapeutic Acceleration Program (Unknown)
Responsible Party: Principal Investigator, Richard Rox Anderson, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2023P003620
Record Dates: First submitted 2024-02-13; First posted 2024-03-08 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Neurofibromas, Cutaneous; Neurofibromatosis 1
MeSH Terms: conditions — Neurofibroma; Neurofibromatosis 1 | interventions — Deoxycholic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treated cutaneous neurofibromas (cNFs) (Active Comparator): Injection into up to 50 cutaneous Neurofibromas (for at total maximum of 10 mL injected) with Kybella (1% deoxycholic acid).
  Interventions: Drug: Kybella
- Control cutaneous neurofibromas (cNFs) (No Intervention): A complementary region of cNFs of similar characteristics to the treatment area in the same body region will be selected to serve as an untreated control group.

INTERVENTIONS:
Drug: Kybella — Kybella is sterile 1% deoxycholic acid provided in a 2 mL single-use vial.
  Other Names: Deoxycholate; Deoxycholic acid
  Arms: Treated cutaneous neurofibromas (cNFs)

SUMMARY:
The goal of this clinical trial is to evaluate the tolerability and effectiveness of multiple treatments of an FDA-approved drug in those with Neurofibromatosis Type 1 (NF1) Cutaneous Neurofibromas (cNFs). The main questions it aims to answer are:

Will performing:

* Up to 6 months treatment sessions
* A minimum of 30 days apart
* With up to 50 injections of deoxycholate into a maximum of 50 cNFs in a single region of the body (for a maximum total dose of 10 mL per monthly treatment session) result in tolerable local skin reactions and reduction in both individual cNF size by >50% as well as improved cNF appearance in the treated field?

Researchers will compare treated tumors and control tumors to see if the treatment is effective.

Participants will:

* Receive up to 6 monthly treatments with Kybella (deoxycholate). Treatment for a given tumor will be stopped when the tumor is assessed as clear clinically.
* Complete surveys asking about pain during and after treatments.
* Complete surveys asking about satisfaction with the treatments.
* Undergo 2D photography and 3D imaging of treatment areas.
* Optionally, receive biopsies of up to 6 treated lesions to investigate characteristics of tumors that respond well to treatment as well as non-respondent tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is an adult ≥18 years of age.
2. Participant has a diagnosis of NF1 based on germline genetic testing or by meeting ≥ 2 the following criteria:

   * Family history of NF1,
   * Six or more light brown ("cafe-au-lait") spots on the skin,
   * Presence of two or more neurofibromas of any type, or one or more plexiform neurofibromas,
   * Freckling under the arms or in the groin area,
   * Two or more pigmented, benign bumps on the eye's iris (Lisch nodules),
   * A distinctive bony lesion: dysplasia (abnormal growth) of the sphenoid bone behind the eye, or dysplasia of long bones, often in the lower leg,
   * Tumor on the optic nerve that may interfere with vision.
3. Participant is seeking treatment for cNF.
4. Participant has ≥ 6 paired cNF that are visible and measure 2 mm or more in size. The target treatment area must be amenable to both deoxycholate injections and surveillance with digital and 3D photography. Preferred locations are trunk (back or chest), arms and legs.
5. Participant is able and willing to comply with all visit, treatment and evaluation schedules and requirements.
6. Participant is able to understand and provide written informed consent.
7. Participant has no known allergy to deoxycholate.
8. Participant has no concurrent injury or wound in the target area.

Exclusion Criteria:

1. Participant cannot give informed consent or adhere to study schedule.
2. Participant is actively tanning during the course of the study.
3. Participant has a known allergy to deoxycholic acid.
4. For female participants: those who are pregnant.
5. Participant has any condition which, in the Investigator's opinion, would make it unsafe (for the participant or study personnel) to treat the participant as part of this research study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 3 months after treatment
  Treatment will be considered tolerable if <40% of participants treated have a >grade 2 CTCAE v5 adverse event (AE).

SECONDARY OUTCOMES:
Patient Reported Outcomes | Baseline, after treatment session #4, and at 3 months after final treatment.
  Using questionnaires we will determine the patients' reported outcomes. Patient Global Assessment: Patient rates degree of change of treated and control cNFs on a scale from -3 (no change) to 3 (very large improvement).
Clinician Reported Outcomes | Baseline, after treatment session #4, and at 3 months after final treatment.
  Using questionnaires we will determine the clinicians' reported outcomes. Physician Global Assessment: Clinician rates degree of change of treated and control cNFs on a scale from -3 (no change) to 3 (very large improvement).
VAS Pain Scale | Baseline, after each treatment session, 1 week after each treatment session, and 3 months after final treatment.
  Participants will be asked to rate their pain using a visual analog scale (0 to 10) at each treatment visit and 1 week post-treatment.
Patient Satisfaction | Baseline, after treatment session #4, and at 3 months after final treatment.
  Satisfaction with each treatment modality is rated from 1 (very unsatisfied) to 5 (very satisfied).
Rate of Healing | Baseline, 1 month, 2 months, 3 months, 4 months, 5 months, 6 months after baseline; 3 months after final treatment.
  Measured clinically via photography completed by a member of the study team at baseline, and all in-person visits.
cNF Appearance (Height) | Baseline, after treatment session #4, and at 3 months after final treatment.
  Clinically completed 2D photography and 3D Cherry Imaging. Change from baseline in height of cNFs.
cNF Appearance (Volume) | Baseline, after treatment session #4, and at 3 months after final treatment.
  Clinically completed 2D photography and 3D Cherry Imaging. Change from baseline in volume of cNFs.

OTHER OUTCOMES:
Biologic Effect/Histology | 3 months after final treatment session.
  A subset of 2-6 cNFs from the treatment region will be assessed after the final treatment session.

CONTACTS AND LOCATIONS:
Overall Officials: Richard R Anderson, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Wellman Center for Photomedicine, Boston, Massachusetts, United States